CLINICAL TRIAL: NCT06690463
Title: Comparison of Diagnostic and Therapeutic Efficacy of Periarticular And/or Intraarticular Lidocaine Injections Under Ultrasound Guidance in Sacroiliac Joint Dysfunction Diagnosis and Treatment
Brief Title: Comparison of Diagnostic and Therapeutic Efficacy of Periarticular And/or Intraarticular Lidocaine Injections Under Ultrasound Guidance in Sacroiliac Joint Dysfunction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jale Zare (Other)
Responsible Party: Sponsor-Investigator, Jale Zare, MD, Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: IstanbulUC-JZare-01
Record Dates: First submitted 2024-11-13; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Sacroiliac Joint Dysfunction; Ultrasound Guided Injection; Intraarticular Injection
Keywords: sacroiliac joint dysfunction, ultrasound guided injection, Periarticular and/or Intraarticular Lidocaine Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Periarticular Lidocaine Injection (Active Comparator): A 2.5 cc injection of 2% lidocaine will be administered to the periarticular area of the sacroiliac joint under ultrasound guidance
  Interventions: Diagnostic Test: sacroiliac joint injection
- Intraarticular Lidocaine Injection (Active Comparator): A 2.5 cc injection of 2% lidocaine will be administered to the articular area of the sacroiliac joint under ultrasound guidance
  Interventions: Diagnostic Test: sacroiliac joint injection
- Periarticular and Intraarticular Lidocaine Injection (Active Comparator): A total 5 cc injection of 2% lidocaine will be administered to the articular and periarticular areas of the sacroiliac joint under ultrasound guidance
  Interventions: Diagnostic Test: sacroiliac joint injection

INTERVENTIONS:
Diagnostic Test: sacroiliac joint injection — The procedure involves the administration of a 2.5 cc injection of 2% lidocaine to the sacroiliac joint, targeting the articular or periarticular areas. The injection is performed under real-time ultrasound guidance to ensure accurate placement of the needle.
  The 2% lidocaine solution is injected into both the joint space (articular area) and the surrounding soft tissues (periarticular area), which may include ligaments, capsules, and adjacent muscles. The goal is to temporarily anesthetize the joint and surrounding structures to assess the contribution of the sacroiliac joint in the patient's pain, as well as to provide therapeutic pain relief. The use of ultrasound ensures minimal risk of injury to surrounding structures and enhances the accuracy of the injection.
  This intervention is commonly used in both diagnostic and therapeutic settings, helping to confirm the role of the sacroiliac joint in a patient's symptoms and providing relief in cases of sacroiliac joint dysfunction.

SUMMARY:
The sacroiliac joint (SIJ) is a joint with unique features, including both hyaline and fibrocartilage, and a discontinuous posterior capsule that enhances stability while minimizing movement. Its innervation is complex and has been a subject of debate, with various studies suggesting that it may be supplied by branches from the lumbosacral plexus, dorsal rami of S1 and S2, and the superior gluteal nerve. Recent studies have confirmed the presence of sensory nerve fibers within the joint capsule and ligaments, indicating that the SI joint is involved in pain and proprioception. Various injury mechanisms, including falls, motor vehicle accidents, and conditions like spondylolisthesis, can lead to SIJ pain. Diagnosis of sacroiliac joint pain involves physical tests, such as the thigh thrust test and compression test, while imaging techniques like scintigraphy have limited value. Provocation tests, particularly when combined, can help identify the source of pain. The primary aim of this study is to evaluate diagnostic interventions for SI joint dysfunction, while secondary aims focus on assessing factors that may affect the quality and generalizability of research on this topic.

DETAILED DESCRIPTION:
The sacroiliac joint is a true diarthrodial joint, surrounded by an articular space containing synovial fluid and encased in a fibrous capsule, but it has unique features not typically found in other diarthrodial joints. The sacroiliac joint contains both hyaline cartilage and fibrocartilage and is characterized by a discontinuous posterior capsule with protrusions and depressions that minimize movement and enhance stability. As a result, the sacroiliac joint is only described as a true synovial joint in its anterior portion. In contrast, the posterior connection, formed by the sacroiliac ligaments, the gluteus medius and minimus muscles, and the piriformis muscle, is a syndesmosis-type joint. The sacroiliac joint is richly equipped with neuro-sensors and proprioceptors. Information regarding its innervation pattern has been a subject of considerable debate. Solonen et al. revealed, based on previous studies, that the innervation of the joint is provided by branches from the lumbosacral plexus, the superior gluteal nerve, the dorsal rami of S1 and S2, and the obturator nerve. However, despite several studies, the exact innervation remains unclear. It has been suggested that the anterior portion is innervated by the sacral plexus, while the posterior portion is innervated by the spinal nerves. It has been proposed that the dominant innervation occurs via the L4-S1 nerve roots, with some contributions from the superior gluteal nerve. Several authors argue that the joint is solely innervated by the sacral dorsal rami. Bernard et al. proposed that the posterior innervation originates from the lateral branches of the posterior rami of L4 to S3, and the anterior innervation is from the region between L2 and S2 segments.

Nakagawa et al. reported that nerve fibers traveling to the sacroiliac joint originate from the ventral rami of L4 and L5, the superior gluteal nerve, and the dorsal rami of L5, S1, and S2. In contrast, Grob and colleagues found that sacroiliac joint innervation is almost entirely derived from the sacral dorsal rami.

Fetal pelvic dissections confirmed that the innervation of the sacroiliac joint originates from the dorsal rami due to the neural fibers being located exclusively in the dorsal mesenchyme.

Murata et al. assessed sensory innervation of the sacroiliac joint in rats and concluded that sensory neurons from the dorsal root ganglia of L1 to S2 on the same side innervate the joint. They also noted that sensory fibers from the L1 and L2 dorsal root ganglia pass through the paravertebral sympathetic chain.

Histological analyses of chronic painful sacroiliac joints have confirmed the presence of nerve fibers within the joint capsule and adjacent ligaments. A recent cadaver study by McGrath and Zhang found that the long posterior sacroiliac ligament received afferent input from S2 in 96% of samples, S3 in 100%, S4 in 59%, and rarely from S1 (4%). Nerve fascicles contained both myelinated and unmyelinated nerve fibers, as well as two morphotypes of paciniform mechanoreceptors and a single non-paciniform mechanoreceptor, suggesting that pain and proprioception may be transmitted through the sacroiliac joint. Szadek et al. concluded that the presence of calcitonin gene-related peptide and substance P immunoreactive fibers in the anterior capsule and interosseous ligaments provides a morphological and physiological basis for pain signals originating from these structures. They also suggested that infiltration techniques used to diagnose sacroiliac joint pain should consider both extra-articular and intra-articular approaches. Sakamoto et al. showed that most mechanoreceptor units in the sacroiliac joint are high-threshold group 3 units, which may have a neuropathic function. However, they argued that proprioceptive function in the sacroiliac joint is limited.

These patterns involve posterior extension to the dorsal sacral foramen, penetration into the L5 epiradicular sheath using the upper space, and ventral leakage into the lumbosacral plexus. Therefore, in the presence of capsular disruption, inflammatory mediators may leak from cracks in the sacroiliac joint into nearby nerve structures and potentially cause radicular pain in some patients.

Several injury mechanisms are associated with the development of sacroiliac joint pain, including direct falls onto the hip, rear-end or lateral motor vehicle accidents, and unexpected situations such as stepping from an uncalculated height or low area. Other identified causes include fusion surgery, anterior lumbar spondylolisthesis, inflammatory and degenerative sacroiliac joint diseases, and many other etiologies.

In a systematic review by Hancock et al., when assessing a range of tests to identify the source of low back pain, including herniated discs, sacroiliac joints, or facet joints, they suggested that a combination of maneuvers that provoke sacroiliac joint pain may be useful in identifying the primary source of symptoms beneath a herniated disc.

A systematic review by Szadek et al. found that the thigh thrust test, compression test, and three or more positive stress tests had sufficient discriminatory power for diagnosing sacroiliac joint pain. A systematic literature review by Song et al. concluded that scintigraphy in patients with ankylosing spondylitis had only limited value in identifying sacroiliitis. A review by Rubinstein and van Tulder, which examined the best evidence for diagnosing neck and low back pain, found moderate evidence for the validity and accuracy of injections. A evidence-based review by Laslett determined that in patients with chronic low back pain, the presence of three or more positive provoked sacroiliac joint tests and the absence of "centralization" were associated with sacroiliac joint pain; this rate was 89% in pregnant women. However, in an evidence-based medicine series by Vanelderen et al., it was concluded that distinguishing sacroiliac joint pain from other types of low back pain based on history and physical examination was difficult. It was also reported that provocation maneuvers had weak predictive value, but the combination of tests could help identify a diagnosis. The primary aim of this review is to systematically evaluate the literature on diagnostic sacroiliac joint interventions. Secondary aims are to analyze factors that may affect the quality and generalizability of the studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 who have signed the volunteer consent form, presenting with complaints of pain radiating to the leg, which may accompany lower back and/or hip pain, and who exhibit tenderness upon palpation consistent with sacroiliac joint involvement, with a positive Fortin finger test.

Exclusion Criteria:

* Injection in the SI joint region (steroid, hyaluronic acid, etc.) in the last 3 months
* History of lumbar (stabilization) and/or hip (prosthesis) surgery
* Presence of inflammatory rheumatic disease
* Evidence of acute or chronic sacroiliitis on imaging
* Active infection in the gluteal area or around the lumbar region (skin, subcutaneous)
* Presence of systemic infectious disease
* Use of anticoagulants that may prevent injection
* Presence of a bleeding disorder
* Uncontrolled diabetes mellitus and/or hypertension
* Pregnancy, lactation
* Presence of psychiatric disorders

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2024-05-22 (Actual); Primary Completion 2024-11-22 (Estimated); Study Completion 2024-12-06 (Estimated)

PRIMARY OUTCOMES:
Pain Relief | Baseline, one hour after injection, one week, and one month
  Pain will be assessed using the Numerical Rating Scale (NRS), which ranges from 0 (no pain) to 10 (worst pain imaginable), during standing, sitting, rising from a chair, walking, lying supine, lying on the painful side, and climbing stairs, both before and after injections into the sacroiliac joint. Higher scores indicate worse pain outcomes.

SECONDARY OUTCOMES:
Overall Improvement | One hour after injection, one week, one month
  Overall improvement will be assessed as a self-reported percentage, ranging from 0% (no improvement) to 100% (complete improvement). Higher percentages indicate better outcomes, with 100% representing full recovery as perceived by the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University - Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murakami E, Tanaka Y, Aizawa T, Ishizuka M, Kokubun S. Effect of periarticular and intraarticular lidocaine injections for sacroiliac joint pain: prospective comparative study. J Orthop Sci. 2007 May;12(3):274-80. doi: 10.1007/s00776-007-1126-1. Epub 2007 May 31. PMID 17530380
- [Background] Kokmeyer DJ, Van der Wurff P, Aufdemkampe G, Fickenscher TC. The reliability of multitest regimens with sacroiliac pain provocation tests. J Manipulative Physiol Ther. 2002 Jan;25(1):42-8. doi: 10.1067/mmt.2002.120418. PMID 11898017
- [Background] Laslett M. Evidence-based diagnosis and treatment of the painful sacroiliac joint. J Man Manip Ther. 2008;16(3):142-52. doi: 10.1179/jmt.2008.16.3.142. PMID 19119403
- [Background] Szadek KM, van der Wurff P, van Tulder MW, Zuurmond WW, Perez RS. Diagnostic validity of criteria for sacroiliac joint pain: a systematic review. J Pain. 2009 Apr;10(4):354-68. doi: 10.1016/j.jpain.2008.09.014. Epub 2008 Dec 19. PMID 19101212
- [Background] Hancock MJ, Maher CG, Latimer J, Spindler MF, McAuley JH, Laslett M, Bogduk N. Systematic review of tests to identify the disc, SIJ or facet joint as the source of low back pain. Eur Spine J. 2007 Oct;16(10):1539-50. doi: 10.1007/s00586-007-0391-1. Epub 2007 Jun 14. PMID 17566796
- [Background] Bowen V, Cassidy JD. Macroscopic and microscopic anatomy of the sacroiliac joint from embryonic life until the eighth decade. Spine (Phila Pa 1976). 1981 Nov-Dec;6(6):620-8. doi: 10.1097/00007632-198111000-00015. PMID 7336283
- [Background] Fortin JD. Sacroiliac Joint DysfunctionA New Perspective. J Back Musculoskelet Rehabil. 1993 Jan 1;3(3):31-43. doi: 10.3233/BMR-1993-3308. PMID 24573095